CLINICAL TRIAL: NCT04262245
Title: Comparison of Different Irrigation Activation Techniques on Postoperative Pain After Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Mustafa Murat Koçak, Associate professor, Bulent Ecevit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-100-04/10
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irrigation activation method (Other): Irrigation activation is a crucial stage of root canal treatment. Therefore, the effect of activation methods on post treatment is an important fact for the comfort of patients.
  Interventions: Procedure: Traditional Irrigation; Device: Xp-endo Finisher (XPF); Device: Passive Ultrasonic Irrigation; Device: EndoActivator

INTERVENTIONS:
Procedure: Traditional Irrigation — irrigation with syringe
Device: Xp-endo Finisher (XPF) — irrigation activation file
Device: Passive Ultrasonic Irrigation — irrigation activation method
Device: EndoActivator — irrigation activation method

SUMMARY:
The aim of this study is to evaluate the effect of different irrigation activation methods on postoperative pain using visual analog scale (VAS) using Xp-endo Finisher, EndoActivator and Passive ultrasonic irrigation activation techniques with traditional irrigation method.

In this study, Traditional Irrigation (GI), Xp-endo Finisher (XPF), Passive Ultrasonic Irrigation (PUI), EndoActivator (EA) techniques will be used for irrigation activation. Twenty-five maxillary or mandibular single root and canal-shaped nonvital teeth will used in each group. Root canals will be prepared with TF-Adaptive system. Four different activation techniques will be applied during final irrigation. The canal treatments will be completed in one stage and postoperative pain analysis will be taken with VAS (Visual Analog Scale) scale after 12-24-48 hours. Statistical analysis will be performed with Mann Whitney-U test.

DETAILED DESCRIPTION:
Vaious irrigation activation techniques have been used endodontic practice. These techniques are used to improve the activity of solutions. The selected techniques in this study are accepted as efficient methods for activation. However, postoperative pan is an important issue for clinicians. Thus, Traditional Irrigation (GI), Xp-endo Finisher (XPF), Passive Ultrasonic Irrigation (PUI), EndoActivator (EA) techniques will be used for irrigation activation. All techniques remove hard and soft tissue remnants successfully. The clinician expect to eliminate the postoperative pain. Therefore, a possible increase in pain due to activation technique may limit the use of these methods. The pain scores will be measured using the scale and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* nonvital tooth
* single rooted tooth

Exclusion Criteria:

* tooth not requiring root canal treatment
* patients under 18 years old
* vital tooth
* tooth having more than 1 canal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative after endodontic treatment | 0-48 hours
  The incidence and severity of pain will be evaluated by using visual analog scale (VAS). The severity of pain varies between 0 to 10, in which 0 means no pain, whislt 10 means unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bülent Ecevit University, Faculty of Dentistry, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No